CLINICAL TRIAL: NCT02102152
Title: Efficacy & Tolerability of Tobramycin Podhaler in Bronchiectasis Patients With Chronic Pseudomonas Aeruginosa Infection
Acronym: TOBI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Mordechai Kremer, Head of Pulmunary Institute, Rabin Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RMCBH147441
Record Dates: First submitted 2014-03-06; First posted 2014-04-02 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-03

CONDITIONS: Bronchiectasis With Chronic Infection With Pseudomonas Aeruginosa
Keywords: Tobramycin Podhaler; bronchiectasis; chronic infection; Pseudomonas Aeruginosa
MeSH Terms: conditions — Bronchiectasis; Persistent Infection; Pseudomonas Infections | interventions — Tobramycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TOBI / Placebo (Active Comparator): TOBI / Placebo.
  Interventions: Drug: Tobramycin
- Placebo / TOBI (Active Comparator): Placebo / TOBI
  Interventions: Drug: Tobramycin

INTERVENTIONS:
Drug: Tobramycin

SUMMARY:
The use of inhaled medications for the treatment of pulmonary diseases allows for the delivery of a high concentration of a drug at the site of disease with reduced systemic absorption and risk of systemic adverse effects. Inhaled Tobramycin has been successfully used in the maintenance treatment of CF patients with chronic colonization with PA (Pseudomonas aeruginosa). In the CF population TOBI has been proven to improve lung functions, decrease the density of the PA in the sputum, decrease hospitalizations, and reduce the risk of mortality.

Non CF Bronchiectasis share many features in common with CF, including frequent colonization with PA that leads to deterioration in lung function and increased morbidity. A recent Cochrane review concluded that there is a small benefit for the use of prolonged antibiotics in the treatment of bronchiectasis, however further randomized controlled trials with adequate power and standardized end points are required.

There have been reports in the literature describing the efficacy of inhaled tobramycin the treatment of patients with non CF bronchiectasis with eradication of PA, and significant improvement in respiratory symptoms. There were however patients who discontinued treatment due to adverse events most commonly cough wheezing and dyspnea. (Scheinberg and Shore, Chest 2005).

TOBI Podhaler is a dry powder inhaler that was recently launched, and is much easier and faster to use compared to nebulised Tobramycin. To the best of our knowledge Tobramycin dry powder formulation has not yet been trialed in patients with non CF bronchiectasis.

The purpose of this trial is to assess the efficacy and tolerability of TOBI Podhaler in patients with non CF bronchiectasis, and to gather more data on the benefit of continuous antibiotic therapy in patients with non CF bronchectais.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with bronchiectasis confirmed by CT
2. Chronic PA colonization with 2 documented sputum cultures positive for PA in the last 24 months.
3. Age >=18

Exclusion Criteria:

1. Patients diagnosed with CF
2. Patients who do not tolerate Tobramycin
3. Pregnant or breastfeeding
4. Patients treated in the last 8 weeks with antibiotic therapy either inhaled or systemic (excluding Azenil PO x 3/week which is allowed)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-04; Primary Completion 2016-04 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Number of exacerbations as measured by number of systemic courses of antibiotics either PO or IV | 52 weeks total
  Exacerbation count at 24 weeks, 48 weeks and 52 weeks

SECONDARY OUTCOMES:
Quality of life and Symptoms Score as measured by SGRQ(Saint George's Respiratory Questionnaire) and CASA-Q-CD (Cough and Sputum Assessment Questionnaire) cough and sputum domains | 52 weeks
  Control Period Patients will visit the site 3 times every 12 weeks, TOBI Period Patients will visit the clinic at least 4 times a year during this 24 week period, when enrolled to the study during the 48 weeks period of the study
Pulmonary function tests (FEV1) | 52 weeks
  Control Period Patients will visit site 3 times every 12 weeks, TOBI Period Patients will visit the clinic at least 4 times a year during this 24 week period, when enrolled to the study during the 48 weeks period of the study
Sputum microbiology: Change in Pseudomona Aeruginosa density in sputum | 52 weeks
  Samples will be taken at every visit and changes will be analyzed at the end of the study, when enrolled to the study during the 48 weeks period of the study PENDING finding a lab that can perform this test (CFU quantitation).
Safety and Tolerability of TOBI podhaler | 52 weeks
  Adverse Events and Serious Adverse Events will be monitored continuously in the study and analyzed at the end of study, when enrolled to the study during the 48 weeks period of the study, plus 4 weeks wash-out.

CONTACTS AND LOCATIONS:
Overall Officials: Mordechai R Kramer, MD, Study Chair — Rabin Medical Center
Locations (1):
- Pulmonary Institute, Rabin Medical Center, Beilinson Campus, Petah Tikva, Israel

REFERENCES:
- [Background] Scheinberg P, Shore E. A pilot study of the safety and efficacy of tobramycin solution for inhalation in patients with severe bronchiectasis. Chest. 2005 Apr;127(4):1420-6. doi: 10.1378/chest.127.4.1420. PMID 15821224
- [Background] Konstan MW, Flume PA, Kappler M, Chiron R, Higgins M, Brockhaus F, Zhang J, Angyalosi G, He E, Geller DE. Safety, efficacy and convenience of tobramycin inhalation powder in cystic fibrosis patients: The EAGER trial. J Cyst Fibros. 2011 Jan;10(1):54-61. doi: 10.1016/j.jcf.2010.10.003. Epub 2010 Nov 12. PMID 21075062
- [Background] Evans DJ, Bara AI, Greenstone M. Prolonged antibiotics for purulent bronchiectasis in children and adults. Cochrane Database Syst Rev. 2007 Apr 18;(2):CD001392. doi: 10.1002/14651858.CD001392.pub2. PMID 17443506